CLINICAL TRIAL: NCT02710578
Title: Acute and Residual Effects of Alcohol on Young Drivers' Performance of Driving Related Skills
Brief Title: Alcohol Effects on Driving-related Skills of Young Drivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Transportation (Unknown)
Responsible Party: Principal Investigator, Robert Mann, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 114/2014
Record Dates: First submitted 2016-02-02; First posted 2016-03-17 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Psychomotor Impairment
Keywords: Alcohol impaired driving; Driving simulation; Residual effects of alcohol; Acute psychomotor effects of alcohol; Young drivers
MeSH Terms: conditions — Psychomotor Disorders | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol (Active Comparator): Alcohol
  Interventions: Drug: Alcohol
- Placebo (Placebo Comparator): Tonic water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alcohol — A single oral administration of an alcoholic beverage mixed in a 1:3 ratio of alcohol (Vodka) to tonic water to obtain a target BAC of 0.08mg%
  Other Names: Smirnoff Vodka
  Arms: Alcohol
Drug: Placebo — A single oral administration of a beverage containing tonic water of the same volume as the alcoholic beverage.
  Other Names: Tonic water
  Arms: Placebo

SUMMARY:
Given the known driving behavior of Driving Under the Influence of Alcohol and some of its parallel to driving under the influence of cannabis, this supplemental study aims to validate the sensitivity of the primary and secondary outcome measures employed in a cannabis and driving study currently in progress.

DETAILED DESCRIPTION:
This study will examine the effects of an intoxicating dose of alcohol on driving-related skills among young drivers using driving simulator technology.

This study is a double-blind, placebo-controlled mixed design study, including randomized between-subjects comparison of the effects of alcohol intoxication and both between- and within-subjects examination of acute and residual effects at approximately 24 and 48 hours following one-time alcohol administration.

Initial contact with potential participants will be made by telephone, where study personnel will conduct a telephone screen for eligibility. Those telephone screened as eligible will attend CAMH for an eligibility assessment. Enrolled participants will complete four sessions on consecutive days: a practice day, an alcohol administration day, and a 24-hour and 48-hour post-alcohol session.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 19 to 25.
* Reported consumption of at least 1 heavy drinking episode (according to NIAAA criteria of 5 drinks for males and 4 for females within an occasion) in the 6 months prior to eligibility assessment.
* Held a valid class G or G2 Ontario driver's license (or equivalent from another jurisdiction) for at least 12 months.
* Willing to abstain from alcohol use for the duration of the study, and for 48 hours prior to Session 2.
* Provides written and informed consent.

Exclusion Criteria:

* Taking medications or have any medical condition for which alcohol is contraindicated
* Is a regular user of medications that affect brain function (i.e., antidepressants, benzodiazepines, stimulants).
* Diagnosis of severe medical or psychiatric conditions.
* Meets criteria for current or lifetime Substance Use Disorders (DSM-IV) with the exception of nicotine.
* Meets criteria for Alcohol Dependence (DSM-IV)
* Is pregnant, is trying to become pregnant, or is currently breastfeeding.
* Severe allergic reaction to citrus.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Psychomotor impairment (driving) | Approximate Time Frame: 30 minutes before, 30 minutes after, 24 and 48 hours after drinking
  The driving simulator will objectively measure changes in driving behaviour after drinking alcohol.

SECONDARY OUTCOMES:
Subjective alcohol effects | Approximate Time Frame: 30 minutes before drinking, 5, 15, 30 minutes and 1, 2, 3, 24 and 48 hours post-drinking
  Visual analogue scale measures how participants feel before and after drinking alcohol. administration.
Cognitive testing | Approximate Time Frame: 30 minutes before drinking, and 1, 24 and 48 hours post-drinking
  Changes in Continuous Performance Test performance.
Breath alcohol content (BAC) | Approximate Time Frame: 30 minutes before drinking, 5, 15, 30, minutes and 1, 2, 3, 24, and 48 hours post-drinking
  Changes in BAC after drinking

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mann, PhD, Principal Investigator — Centre for Addiction and Mental Health; Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health; Bruna Brands, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lenne MG, Dietze PM, Triggs TJ, Walmsley S, Murphy B, Redman JR. The effects of cannabis and alcohol on simulated arterial driving: Influences of driving experience and task demand. Accid Anal Prev. 2010 May;42(3):859-66. doi: 10.1016/j.aap.2009.04.021. PMID 20380913
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research